CLINICAL TRIAL: NCT04326764
Title: A Randomized, Multicenter Phase III Study to Assess the Efficacy of Panobinostat Maintenance Therapy vs. Standard of Care Following Allogeneic Stem Cell Transplantation in Patients With High-risk AML or MDS (ETAL-4 / HOVON-145)
Brief Title: Panobinostat Maintenance After HSCT fo High-risk AML and MDS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change of marketing authorisation holder
Sponsor: Goethe University (Other)
Collaborators: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other); Polish Adult Leukemia Group (Other); Schweizerische Arbeitsgemeinschaft für klinische Krebsforschung (Unknown)
Responsible Party: Principal Investigator, Gesine Bug, Director of Transplant Program, Principal Investigator, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETAL-4 / HOVON-145
Record Dates: First submitted 2019-03-21; First posted 2020-03-30 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukaemia (AML); Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Panobinostat (Experimental): Panobinostat 20 mg oral three times weekly every second week
  Interventions: Drug: Panobinostat
- Standard of Care (No Intervention): Treatment according to local standards

INTERVENTIONS:
Drug: Panobinostat — Panobinostat should be taken orally once on each scheduled day at about the same time, either with or without food. Each dose of panobinostat should be taken with a cup of water.
  The capsules should be swallowed as whole. If vomiting occurs during the course of treatment, no re-dosing is allowed before the next scheduled dose. If one dose is forgotten during the morning on a scheduled treatment day then the missed dose should be taken on that same day within 12 hours. After more than 12 hours, that day's dose should be withheld, and the patient should wait to take panobinostat until the next schedule treatment day. The patient should then continue treatment with the original dosing schedule.
  Panobinostat will be administered at a dose of 20 mg three times weekly (TIW) every second week and will be dosed on a flat scale of mg/day and not by weight or body surface area.
  Panobinostat will be dispensed as a 20 mg capsule or as two 10 mg capsules.
  Other Names: Farydak
  Arms: Panobinostat

SUMMARY:
Aim of this prospective randomized trial is to compare maintenance treatment with panobinostat interspersed with donor lymphocyte infusions (DLI) versus the standard approach of pre-emptive DLI alone in patients with poor-risk AML/MDS having favorably received an allogeneic HSCT followed by engraftment, donor chimerism and hematopoietic reconstitution.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) has been shown to improve the outcome of poor-risk AML and MDS in both younger and older patients. Reduced-intensity conditioning (RIC) regimen have partially abrogated the problem of regimen-related toxicity. However, graft-versus-host disease (GvHD) remains a major cause of non-relapse morbidity and mortality. Despite a strong graft versus leukemia (GvL) effect after allogeneic HSCT, the relapse rate after transplantation in poor-risk leukemia patients is still too high, necessitating new approaches to exploit GvL in a more optimized way. In addition, minimizing the GvHD reaction remains an important goal. One attractive strategy may be the administration of epigenetic therapy early after HSCT in order to optimize the GvL effect, to provide a direct anti-leukemic effect, and to control GvHD. Two preceding phase I/II studies have suggested that post-transplant administration of the histone deacetylase (HDAC) inhibitor panobinostat may be associated with a reduced relapse rate, while allowing for control of GvHD. Based on these two studies, the hypothesis of the present trial is that panobinostat can be an effective drug in preventing relapse by optimizing GvL in MDS and AML patients with high-risk features after HSCT, while at the same time reducing GvHD. It has been designed to test this hypothesis in a prospective randomized trial comparing maintenance with panobinostat interspersed with donor lymphocyte infusions (DLI) versus the standard approach of pre-emptive DLI alone in patients with poor-risk AML/MDS having favorably received an allogeneic HSCT followed by engraftment, donor chimerism and hematopoietic reconstitution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-70 years of age)
* AML (except acute promyelocytic leukemia with PML-RARA and AML with BCR-ABL1) according to WHO 2016 classification with high-risk features defined as one or more of the following criteria:

  * refractory to or relapsed after at least one cycle of standard chemotherapy
  * > 10% bone marrow blasts at day 14-21 of the first induction cycle
  * adverse risk according to ELN 2017 risk stratification by genetics (Appendix 2) regardless of stage
  * secondary to MDS or radio-/chemotherapy
  * MRD positive before HSCT based on flow cytometry or PCR

or

* MDS with excess blasts (MDS-EB) according to the WHO 2016 classification, or high-risk or very high-risk according to IPSS-R

and

First allogeneic HSCT scheduled within the next 4-6 weeks using one of the following donors, conditioning regimens and strategies for GvHD prophylaxis:

1. Matched sibling or matched unrelated donor (i.e. 10/10 or 9/10 HLA-matched) or haploidentical family donor
2. Conditioning regimens:

   1. Reduced-intensity conditioning:

a. Fludarabine/Melphalan b. Fludarabine/Busulfan2 (FB2) (2) Myeloablative conditioning:

1. Fludarabine/Busulfan4 (FB4)
2. Busulfan/Cyclophosphamide (BU/CY)
3. Fludarabine/TBI 8 Gy
4. Cyclophosphamide/TBI 12 Gy (3) Fludarabine/Cyclophosphamide/TBI 2 Gy in combination with post-Tx cyclophosphamide (TP-CY) only (4) Thiotepa/Busulfan/Fludarabine (TBF) in the context of an haploidentical HSCT only (5) In case of active disease at HSCT, salvage chemotherapy prior to conditioning is permitted

c. Strategies for GvHD prophylaxis:

1. HLA-matched donors:

   a. CSA + MMF +/- ATG b. CSA + MTX +/- ATG c. PT-CY + CSA
2. Haploidentical donors:

   d. PT-CY + CSA + MMF

   - No history of significant cardiac disease and absence of active symptoms, otherwise documented left ventricular EF ≥ 40%

   - Written informed consent for registration

   Exclusion Criteria:

   - Prior treatment with a DAC inhibitor

   - Hypersensitivity to the active substance or to any of the excipients of panobinostat
   * HIV or HCV antibody positive
   * Psychiatric disorder that interferes with ability to understand the study and give informed consent, and/or impacts study participation or follow-up.
   * Female patients who are pregnant or breast feeding
   * History of another primary malignancy that is currently clinically significant or currently requires active intervention

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
  OS is measured from date of randomization to the date of death or date of last follow up. Observations of patients alive at last follow up will be censored at date of last follow up.

SECONDARY OUTCOMES:
Event-free survival (EFS) | 5 years
  EFS is defined as time interval from randomization until relapse of MDS or AML, any treatment of molecular relapse (except DLI) or death from any cause, whichever occurs first. Observations of patients without any event will be censored at time of last follow up.
Disease-free survival (DFS) | 5 years
  DFS is defined as time interval from randomization until relapse of MDS or AML, or death from any cause, whichever occurs first. Observations of patients without any event will be censored at time of last follow up.
Cumulative incidence of hematologic relapse | 5 years
  Remission duration is defined as time from randomization until relapse (including any treatment (except DLI) of molecular relapse). Death in complete remissions (CR) is considered as competing event for relapse. Patients for whom no relapse nor death in CR was observed will be censored at date of last follow up.
Cumulative incidence, time and cause of non-relapse mortality (NRM) | 5 years
  Time to NRM is defined as time from randomization until death in CR from any cause. Relapse is considered as competing event for NRM. Patients for whom no death in CR nor relapse was observed will be censored at date of last follow up.
Cumulative incidence of new onset or aggravation of acute GvHD grade III-IV | 5 years
  Cumulative incidence of new onset or aggravation acute GvHD grade III-IV is calculated as number of patients who newly experienced acute GvHD grade III-IV after randomization or whose preexisting lower grade acute GvHD aggravated to grade 3 or 4 divided by all patients in the analysis set. Cumulative incidence is calculated separately for each arm.
Cumulative incidence and maximal grade of severity of chronic GvHD requiring systemic treatment within one year after HSCT | 1 year
  Acute and chronic GvHD will be graded according to NIH consensus criteria. In case of chronic GvHD, evaluation forms provided by the NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host-Disease should be used.
  Time to chronic GvHD requiring systemic treatment is defined time from randomization until date of first diagnosis of chronic GvHD requiring systemic treatment. Relapse and death in CR without chronic GvHD requiring systemic treatment are considered as competing events. Patients for whom no chronic GvHD, nor relapse, nor death in CR was observed will be censored at date of last follow up.
Percentage of patients who are free of systemic immunosuppressive therapy at one and two years after HSCT | 2 years
  Percentage of patients who are free of systemic immunosuppressive therapy is calculated as number of patients who are free of systemic immunosuppressive therapy at the respective time point divided by the total number of patients in the analysis set multiplied by 100. The percentage is calculated separately for each arm.
Percentage of patients completing the one year study treatment and duration of panobinostat administration in patients who discontinue study treatment prematurely | 1 year
  Percentage of patients completing the one year study treatment is calculated as number of patients completing the one year study treatment divided by the total number of patients in the analysis set multiplied by 100. The percentage is calculated for the panobinostat arm only.
  The duration of panobinostat administration is calculated from date of first administered dose of study medication until date of last administered dose of study medication.
Percentage of patients with minimal residual disease (MRD) conversion from baseline to 6 months after HSCT | 6 months
  Percentage of patients with MRD conversion from baseline to 6 months after HSCT is calculated as number of patients who were MRD positive at baseline and are MRD negative at 6 months after HSCT divided by the number of patients who were MRD positive at baseline.
  Patients who were MRD negative at baseline will not be considered in this endpoint.
Patient-reported HRQoL during panobinostat maintenance therapy | 4 years
  Patient reported health-related quality of life will be assessed using the cancer generic 'European Organization for Research and Treatment of Cancer' quality of life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gesine Bug, PD Dr., Principal Investigator — Goethe University Frankfurt
Locations (19):
- Germany (14):
  - Robert Bosch Krankenhaus, Stuttgart, Baden-Wurttemberg
  - University Hospital Jena, Jena, Thuringia
  - Universitätsklinikum Leipzig, Leipzig, Thuringia
  - Klinikum Augsburg, Augsburg
  - University Hospital Bonn, Bonn
  - Universtity Hospital Dresden, Dresden
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Otto-von-Guericke University, Magdeburg
  - Universitätsmedizin Mainz, Mainz
  - Klinikum Mannheim, Mannheim
  - Philipps-Universität Marburg, Marburg
  - University Hospital Münster, Münster
  - Klinikum Nürnberg Nord, Nuremberg
- Netherlands (5):
  - Amsterdam University Medical Center - VUMC, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht
  - Radboud UMC, Nijmegen
  - Erasmus University Medical Center, Rotterdam